CLINICAL TRIAL: NCT00610740
Title: WCC# 44: A Pilot Study of CerviPrep, a Novel Drug Delivery Device for the Cervix, in the Local Administration of Gemcitabine, a Radiation Sensitizer
Brief Title: CerviPrep for Applying Topical Gemcitabine to the Cervix in Treating Patients With Primary Endometrial, Cervical, or Ovarian Epithelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005LS071; WCC #44 (Other: Women's Cancer Center, University of Minnesota); UMN-0510M6486 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-02-07; First posted 2008-02-08 (Estimated); Results first posted 2010-06-17 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Cervical Cancer; Endometrial Cancer; Ovarian Cancer
Keywords: recurrent cervical cancer; cervical cancer; endometrial carcinoma; ovarian epithelial cancer; recurrent ovarian epithelial cancer; recurrent endometrial carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Gemcitabine; Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients Treated with CerviPrep™ (Experimental): CerviPrep™, a novel drug delivery device, was developed specifically for applying pharmaceuticals directly on the cervix. It consists of a syringe-like tube attached to a plastic cap that covers the cervix. Drug can be delivered through the tube, directly to the cervix without spillage onto vaginal or vulvar tissues.
  Interventions: Drug: topical gemcitabine hydrochloride; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: topical gemcitabine hydrochloride — Gemcitabine 100 mg/m2 will be administered as a single dose, directly to the cervix via the CerviPrep™ device.
  Other Names: Gemzar
Procedure: therapeutic conventional surgery — hysterectomy
  Other Names: removal of uterus

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Using the CerviPrep™ drug delivery device to apply topical gemcitabine to the cervix may be an effective way to kill more tumor cells.

PURPOSE: This phase II trial is studying how well CerviPrep™ works in applying topical gemcitabine to the cervix in treating patients with primary endometrial cancer, cervical cancer, or ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of the CerviPrep™ device in delivering topical gemcitabine hydrochloride to the cervix

Secondary

* To document any side effects directly attributed to local administration of gemcitabine hydrochloride.

OUTLINE: Patients undergo application of topical gemcitabine hydrochloride directly to the cervix using the CerviPrep™ drug delivery device during routine hysterectomy.

Uterine vein and peripheral blood samples are obtained periodically to measure local and peripheral gemcitabine hydrochloride concentration levels in the blood. Local gemcitabine hydrochloride concentration levels are also measured in uterine tissue samples obtained from the surgical specimen after hysterectomy.

Patients complete a self-reported symptom diary for the first 7 days after surgery for assessment of local and systemic side effects associated with topical administration of gemcitabine hydrochloride.

After completion of study therapy, patients are followed at 2-4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary endometrial or cervical cancer
* Scheduled to undergo abdominal hysterectomy as part of surgical staging and/or treatment
* Gynecologic Oncology Group (GOG) performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm³
* Platelet count ≥ 100,000 cells/mm³
* Creatinine ≤ 2.5 mg/dL
* Serum Aspartate aminotransferase (AST) or Alanine transaminase (ALT) ≤ 3 times upper limit of normal
* Total bilirubin ≤ 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion Criteria:

* Serious medical condition or psychiatric illness that places the patient at an unacceptable risk for study participation or precludes signing the informed consent
* Known allergic reaction or hypersensitivity to gemcitabine hydrochloride
* Prior radiotherapy to the whole abdomen or pelvis
* More than 28 days since prior standard or experimental anticancer therapy
* No other concurrent anticancer agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Levi S. Downs, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 additional patients were consented, but never treated.
Groups:
- Patients Treated With CerviPrep™: During routine hysterectomy for endometrial or cervical carcinoma apply topical gemcitabine 100mg/m^2 using CerviPrep™ drug delivery system. CerviPrep™, a novel drug delivery device, was developed specifically for applying pharmaceuticals directly on the cervix. It consists of a syringe-like tube attached to a plastic cap that covers the cervix. Drug can be delivered through the tube, directly to the cervix without spillage onto vaginal or vulvar tissues.
Period: Overall Study
Arm/Group | Patients Treated With CerviPrep™
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Treated With CerviPrep™
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] — All 23 patients are included in this measure - only 18 participated and were treated.
  Years | 50.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Measurable Concentration of Gemcitabine in Uterine Vein (dFdC)
Description: Efficacy of the CerviPrep™ device in delivering topical gemcitabine hydrochloride to the cervix as measured by gemcitabine hydrochloride concentration levels in tissue samples.
Time Frame: 30 Minutes After Application of Gemcitabine
Measure: Number; unit: Participants
Arm/Group | Patients Treated With CerviPrep™
Number analyzed (Participants) | 18
Participants | 5 (8.2)

2. Primary Outcome: Number of Patients With Measurable Concentration of Gemcitabine Metabolites in Uterine Vein (dFdU)
Description: Efficacy of the CerviPrep™ device in delivering topical gemcitabine hydrochloride to the cervix as measured by local (uterine vein) gemcitabine hydrochloride concentration levels in blood
Time Frame: 30 minutes post administration
Measure: Number; unit: Participants
Arm/Group | Patients Treated With CerviPrep™
Number analyzed (Participants) | 18
Participants | 3 (80.7)

3. Secondary Outcome: Number of Patients With Measurable Peripheral Vein Concentration of dFdC
Description: Efficacy of the CerviPrep™ device in delivering topical gemcitabine hydrochloride to the cervix as measured by peripheral gemcitabine hydrochloride concentration levels in blood
Time Frame: 30, 60, 90 minutes post uterine vein sample
Measure: Number; unit: Participants
Arm/Group | Patients Treated With CerviPrep™
Number analyzed (Participants) | 18
Participants
  30 Minutes | 0
  60 Minutes | 0
  90 Minutes | 0

ADVERSE EVENTS:
Time Frame: Day 1 of treatment through 30 Days post treatment
Arm/Group | Patients Treated With CerviPrep™
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With CerviPrep™ (N=18)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes